CLINICAL TRIAL: NCT05762523
Title: An Open-label Controlled Study of the Safety and Tolerability of the Live Cell-based Vaccine Against Smallpox and Other Orthopoxvirus Infections (VAC∆6 Vaccine) Based on Vaccinia Virus, in Volunteers Aged 18-40 Years
Brief Title: Safety and Tolerability Study of the VAC∆6 Vaccine in Volunteers Aged 18-40 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal Budgetary Research Institution State Research Center of Virology and Biotechnology "Vector" (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC∆6-01/18
Record Dates: First submitted 2023-01-23; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Smallpox; Monkeypox; Cowpox; Vaccinia Virus Infection
Keywords: VAC∆6 vaccine; Smallpox; Оrthopoxviruses; Сlinical study
MeSH Terms: conditions — Smallpox; Mpox, Monkeypox; Cowpox | interventions — Smallpox Vaccine

STUDY DESIGN:
Intervention Model Description: This study is an open-label, controlled, parallel-group clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 "VAC∆6: оnce at a dose of 10⁶ PFU (plaque-forming units)" (Experimental): 15 healthy volunteers of both sexes aged 18-40 years who had not been vaccinated against smallpox, had no vaccine marks and anti-smallpox virus neutralizing antibodies in their sera as well as those who met the inclusion criteria and did not have any exclusion criteria
  Interventions: Biological: VAC∆6 vaccine - оnce at a dose of 10⁶ PFU
- Group 2 "VAC∆6: once at a dose of 10⁷ PFU" (Experimental): 15 healthy volunteers of both sexes aged 18-40 years who had not been vaccinated against smallpox, had no vaccine marks and anti-smallpox virus neutralizing antibodies in their sera as well as those who met the inclusion criteria and did not have any exclusion criteria
  Interventions: Biological: VAC∆6 vaccine - once at a dose of 10⁷ PFU
- Group 3 "VAC∆6: twice at a dose of 10⁶ PFU" (Experimental): 15 healthy volunteers of both sexes aged 18-40 years who had not been vaccinated against smallpox, had no vaccine marks and anti-smallpox virus neutralizing antibodies in their sera as well as those who met the inclusion criteria and did not have any exclusion criteria
  Interventions: Biological: VAC∆6 vaccine - twice at a dose of 10⁶ PFU
- Group 4 "OspaVir® + live smallpox vaccine" (Experimental): 15 healthy volunteers of both sexes aged 18-40 years who had not been vaccinated against smallpox, had no vaccine marks and anti-smallpox virus neutralizing antibodies in their sera as well as those who met the inclusion criteria and did not have any exclusion criteria
  Interventions: Biological: Live smallpox vaccine (Smallpox vaccine) + The OspaVir® inactivated smallpox vaccine

INTERVENTIONS:
Biological: VAC∆6 vaccine - оnce at a dose of 10⁶ PFU — 15 volunteers vaccinated once intradermally at a dose of 10⁶ PFU (0.2 ml) of the VAC∆6 vaccine in the outer surface of the shoulder 8-10 cm below the shoulder joint
  Arms: Group 1 "VAC∆6: оnce at a dose of 10⁶ PFU (plaque-forming units)"
Biological: VAC∆6 vaccine - once at a dose of 10⁷ PFU — 15 volunteers vaccinated once intradermally at a dose of 10⁷ PFU (0.2 ml) of the VAC∆6 vaccine in the outer surface of the shoulder 8-10 cm below the shoulder joint
  Arms: Group 2 "VAC∆6: once at a dose of 10⁷ PFU"
Biological: VAC∆6 vaccine - twice at a dose of 10⁶ PFU — 15 volunteers vaccinated twice spaced 28 days apart, intradermally at a dose of 10⁶ PFU (0.2 ml) of the VAC∆6 vaccine in the outer surface of the shoulder 8-10 cm below the shoulder joint
  Arms: Group 3 "VAC∆6: twice at a dose of 10⁶ PFU"
Biological: Live smallpox vaccine (Smallpox vaccine) + The OspaVir® inactivated smallpox vaccine — 15 volunteers vaccinated by the two-step vaccination method: Step 1 - the first vaccination once subcutaneously with 1 dose (0.5 ml) of the inactivated smallpox vaccine OspaVir® in the area of the left shoulder 8-10 cm below the shoulder joint; Step 2 - the second vaccination once by the method of multiple puncture into the outer surface of the shoulder 8-10 cm below the shoulder joint with a live smallpox vaccine at a dose of 1x 106 PFU 7 days following the first vaccination with OspaVir®.
  Arms: Group 4 "OspaVir® + live smallpox vaccine"

SUMMARY:
The aim of the clinical study is to study the safety and tolerability of the live cell-based vaccine against smallpox and other orthopoxvirus infections (VAC∆6 vaccine) based on vaccinia virus, in intracutaneous administration.

The research tasks are to:

* evaluate the safety of various schemes for the use of the VAC∆6 vaccine using a set of clinical and laboratory-instrumental methods (thermometry, blood pressure registration, auscultation of the heart and lungs, electrocardiography (ECG), complete blood count and common urine test, biochemical, immunological, and virological studies);
* evaluate the reactogenicity of various schemes for the use of the VAC∆6 vaccine (taking into account the number of local and systemic reactions, the percentage of those vaccinated with various degrees of manifestation of systemic and local reactions);
* evaluate the possibility of virus shedding into the environment by volunteers;
* evaluate the immunological efficacy of various vaccine administration schemes;
* identify the development of undesirable reactions to the administration of the vaccine;
* evaluate the cellular immune response to the introduction of various schemes for the use of the vaccine;
* evaluate preliminary efficacy data in order to select an optimal scheme for the administration of the vaccine to make a decision on conducting Phase II clinical trials in an extended group of volunteers.

DETAILED DESCRIPTION:
This study is an open-label, controlled, parallel-group clinical trial. The study included 60 healthy volunteers of both sexes aged 18-40 years who had not been vaccinated against smallpox, had no vaccine marks and anti-smallpox virus neutralizing antibodies in their sera as well as those who met the inclusion criteria and did not have any exclusion criteria.

Distribution of volunteers by groups:

Group 1: 15 volunteers vaccinated once intradermally at a dose of 10⁶ plaque-forming units (PFU) (0.2 ml) of the VAC∆6 vaccine in the outer surface of the shoulder 8-10 cm below the shoulder joint; Group 2: 15 volunteers vaccinated once intradermally at a dose of 10⁷ PFU (0.2 ml) of the VAC∆6 vaccine in the outer surface of the shoulder 8-10 cm below the shoulder joint; Group 3: 15 volunteers vaccinated twice spaced 28 days apart, intradermally at a dose of 10⁶ PFU (0.2 ml) of the VAC∆6 vaccine in the outer surface of the shoulder 8-10 cm below the shoulder joint; Group 4: 15 volunteers vaccinated by the two-step vaccination method: Step 1 - the first vaccination once subcutaneously with 1 dose (0.5 ml) of the inactivated smallpox vaccine OspaVir® in the area of the left shoulder 8-10 cm below the shoulder joint; Step 2 - the second vaccination once by the method of multiple puncture into the outer surface of the shoulder 8-10 cm below the shoulder joint with a live smallpox vaccine at a dose of 1x 10⁶ PFU 7 days following the first vaccination with OspaVir®.

Since the product "Live cell-based vaccine against smallpox and other orthopoxvirus infections (VAC∆6 vaccine) based on vaccinia virus" was used for the first time for human vaccination, the vaccination of volunteers was started at a low dose, i.e. 1x10⁶ PFU.

The first five volunteers included in Group 1 were vaccinated intradermally at a dose of 1x10⁶ PFU. The volunteers were monitored daily; 14 days after vaccination, in the absence of side effects and after the results were agreed upon, vaccination was performed for the remaining 10 Group 1 volunteers and the first 5 volunteers of Group 2 who were vaccinated at a dose of 1x10⁷ PFU. After 14 days, in the absence of adverse effects (AEs) or serious adverse effects (SAEs), the rest of the volunteers included in Group 2 were vaccinated.

After receiving the results indicating the absence of AEs or SAEs in the volunteers vaccinated once with the VAC∆6 vaccine at a dose of 1x10⁶ PFU, the first vaccination of Group 3 volunteers was performed, the dose of the vaccine was 1x10⁶ PFU, and after 28 days - the second vaccination was performed.

Group 4 was vaccinated with reference products: live smallpox vaccine (smallpox vaccine) and the OspaVir® vaccine, an inactivated smallpox vaccine.

Vaccination was performed in two steps:

* the first step: subcutaneous administration of the inactivated smallpox vaccine OspaVir®;
* the second step: skin inoculation with a live smallpox vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate in the study after written informing.
2. Healthy volunteers (men and women) aged 18 to 40:

   * absence of somatic or infectious diseases during the last 6 months;
   * body weight of volunteers should not go beyond 20% of the ideal body weight for a given sex, age, and height;
   * absence during the last 6 months of antiviral therapy, the use of steroids (except for the local use of steroids in the form of ointments, eye drops, sprays or inhalations), immunomodulatory dugs;
   * persons not infected with HIV, viral hepatitis B and C, lues;
   * clinical and laboratory parameters within the range as follows: leukocytes: from 4,000 to 10,000 cells/mm³; platelets: 180,000 to 320,000 per mm³.

Exclusion Criteria:

1. Hypersensitivity to any component of the product, allergy to vaccine components.
2. Pregnancy or breastfeeding.
3. The military.
4. Persons in custody in detention facilities and those serving sentences in correctional facilities.
5. Children under the age of 18.
6. Acute infectious or non-infectious diseases, exacerbation of chronic diseases less than 4 weeks prior to the study.
7. Tuberculosis (pulmonary and extrapulmonary).
8. Skin diseases: a) common dermatoses (pemphigus, psoriasis, eczema, atopic dermatitis), including those in the past; other acute and chronic diseases or impaired skin cover (burns, impetigo, herpes, herpes zoster chicken pox, pustular diseases).
9. Immunosuppressive conditions: congenital or acquired immunodeficiency syndrome (including HIV infection), leukemia, malignant neoplasms, organ transplantation, cellular and humoral immunodeficiencies.
10. Immunosuppressive therapy: treatment with antimetabolites, high doses of corticosteroids for 14 days or more, radio and x-ray therapy, etc.
11. Cardiovascular diseases: decompensated heart defects, subacute bacterial endocarditis, myocarditis, pericarditis, hypertension of II-III degrees, angina pectoris, myocardial infarction; other forms of pathology: hypertension of the 1st degree, well-controlled heart defects, angina pectoris (mild forms).
12. Diseases of the kidneys and urinary tract: diffuse glomerulonephritis, congenital nephropathy, chronic renal failure, pyelonephritis, toxic nephropathy (transient).
13. Diseases of the digestive system: cirrhosis of the liver, chronic hepatitis, hepatocerebral dystrophy, acute and chronic pancreatitis, diseases of the biliary tract, gastric ulcer and duodenal ulcer, ulcerative colitis.
14. Diseases of the endocrine system: diabetes mellitus, severe forms of thyrotoxicosis and adrenal insufficiency or dysfunction, thymomegaly, congenital enzymopathy.
15. Systemic connective tissue diseases: systemic lupus erythematosus, discoid lupus, rheumatism, rheumatoid arthritis, systemic vasculitis, systemic scleroderma.
16. Blood diseases: leukemia, Hodgkin's disease, aplastic anemia, hemophilia, Werlhof's disease; hemolytic conditions; deficiency anemia.
17. Allergic diseases: bronchial asthma; asthmatic bronchitis, asthmatic syndrome (associated with a respiratory infection); severe anaphylactic reactions (shock, angioedema of the larynx, etc.) to a variety of food, drug and other allergens; allergic reactions to individual allergens (various rashes, clinical disorders, etc.).
18. Diseases of the ear, throat, nose: chronic tonsillitis and adenoiditis requiring surgical treatment; chronic otitis.
19. Surgery within the previous 2 months.
20. Simultaneous participation in other clinical trials.
21. Persons with alcohol, drug or drug addiction.
22. The presence of mental illness and neurasthenia.
23. Previous treatment with human immunoglobulin preparations, if less than 6 months have passed since the treatment.
24. Failure to meet inclusion criteria.
25. Vaccination with any vaccine less than 2 months prior to study entry.
26. Premenopausal women (last menstrual period ≤ 1 year prior to signing the informed consent) who are not surgically sterile.
27. Women who have reproductive potential or do not use or plan to use approved birth control products throughout the study nor they agree to a urine pregnancy test while participating in the study. Acceptable birth control methods include extrauterine devices, oral, implanted, or injectable contraceptives.
28. Nervous and mental diseases: injuries of the central nervous system (CNS) with residual effects, encephalitis and encephalomyelitis (including post-vaccination), meningitis, polyradiculoneuritis (including those in the past), epilepsy, decompensates or subcompensated hydrocephalus, demyelinating and degenerative lesions of the nervous system (muscle degeneration, etc.), stroke; compensated hydrocephalus, Down's disease, Little's disease, CNS trauma without residual effects, history of febrile convulsions, mental illness.
29. Positive analysis for HIV, viral hepatitis B and C, lues.
30. Concomitant diseases that, in the opinion of the investigator, may interfere with the evaluation of the objectives of the study.
31. Serious post-vaccination reactions/complications associated with any previous vaccination.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-18 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Changes in the percentage of vaccinees with a titer of virus-neutralizing antibodies to vaccinia virus ≥1:40, at specified time intervals. | Groups 1, 2, 3: at days 0, 21, 30, 60, 90, 180. Group 4: at days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, the percentage of the vaccinees with a titer of virus-neutralizing antibodies to vaccinia virus ≥1:40 is recorded in the neutralization test in embryonated chicken eggs.
  Value changes of this indicator between time points are assessed.
Recording the number of local reactions. | Groups 1, 2: at days 0 - 14, 21. Group 3: at days 0 - 14, 21, 28 - 42, 49. Group 4: at days 0 - 22, 29.
  On control days, the sum of local reactions is recorded: formation of inoculation elements (redness, swelling and papulo-nodules, pustules, vesicles, erythema, induration). Value changes of this indicator between time points are assessed.
  Evaluation criteria for local reactions:
  1. The intensity or severity of adverse reactions should be assessed on a 4-point scale: 0 - none (no symptoms); 1 - mild (presence of mild symptoms); 2 - medium (symptoms that noticeably impair normal daily activities); 3 - severe (symptoms that interfere with normal daily activities).
  2. The severity of local reactions was assessed according to the following criteria:
     * Hyperemia < 50.0 mm (⌀) or an infiltrate < 25.0 mm (⌀) - weak;
     * Hyperemia ≤ 50.0 mm (⌀) or an infiltrate 26.0-50.0 mm (⌀) - medium;
     * Infiltrate > 50.0 mm (⌀) - strong.

SECONDARY OUTCOMES:
Changes in the activity of delayed-type hypersensitivity (DTH) effectors to vaccinia virus at specified time intervals. | Groups 1, 2: at days 1, 30, 90. Groups 3, 4: at days 1, 30, 60, 90.
  On control days, the changes in the activity of DTH effectors to vaccinia virus are assessed. The assessment of the activity of specific DTH effectors in vitro should be carried out according to the migration index (MI), which characterizes the migration activity of leukocytes; according to the migration inhibition index (MII), which characterizes the intensity of lymphokine production, and according to the integral indicator of the effector functions (IEF). The reaction is considered positive if the difference between the experimental and control values is greater than 20%.
Changes in the content of Class A, M, G, and E immunoglobulins. | Groups 1, 2, 3: at days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: at days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, the changes in the content of Class A (in mg/ml), M (in mg/ml), G (in mg/ml), and E (in IU/ml) immunoglobulins is assessed.
Changes in the content of T cells and their subpopulations: cluster of differentiation 3 (CD3+), cluster of differentiation 4 (CD4+), cluster of differentiation 8 (CD8+), CD4+/CD8+. | Groups 1, 2, 3: at days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: at days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, the changes in the content of T cells and their subpopulations is assessed: CD3+ (in % in relation to the total number of lymphocytes), CD4+ (in % in relation to CD3+), CD8+ (in % in relation to CD3+), CD4+/CD8+.
Recording the number of systemic reactions. | Groups 1, 2: at days 0 - 14, 21. Group 3: at days 0 - 14, 21, 28 - 42, 49. Group 4: at days 0 - 22, 29.
  Recording the number of systemic reactions (malaise, headache, rise in body temperature, weakness, sweating, sleep and appetite disorders, nausea, vomiting, abdominal pain, etc.). Evaluating criteria for systemic reactions:
  1. The intensity or severity of adverse reactions should be assessed on a 4-point scale: 0 - none (no symptoms); 1 - mild (presence of mild symptoms); 2 - medium (symptoms that noticeably impair normal daily activities); 3 - severe (symptoms that interfere with normal daily activities).
  2. The temperature response should be evaluated according to the following categories in °С: 0 (none) ≤ 37 °C; 1 (weak) > 37 °С - ≤ 37.5 °С; 2 (medium) > 37.5 °С - ≤ 38.5 °С; 3 (strong) > 38.5°C.
Recording of the percentage of the vaccinated with various degrees of manifestation of systemic and local reactions. | Groups 1, 2: at days 0 - 14, 21. Group 3: at days 0 - 14, 21, 28 - 42, 49. Group 4: at days 0 - 22, 29.
  Recording of the percentage of the vaccinated with various degrees of manifestation of systemic and local reactions.

OTHER OUTCOMES:
Body temperature monitoring at specified time intervals. | Groups 1, 2, 3: at days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: at days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  Body temperature is recorded (in degrees Celsius, °C) on control days. The changes in the values of this indicator between time points are assessed.
Arterial blood pressure monitoring at specified time intervals. | roups 1, 2, 3: at days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: at days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  Systolic and diastolic blood pressure is recorded (in mmHg). The changes in the values of this indicator between time points are assessed.
Heart rate monitoring at specified time intervals. | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  The heart rate is recorded (in beats per minute) on control days. The changes in the values of this indicator between time points are assessed.
Monitoring of the frequency of respiratory movements at specified time intervals. | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.]
  The frequency of respiratory movements (per minute) is recorded on control days. The changes in the values of this indicator between time points are assessed.
Monitoring of the content of erythrocytes (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of erythrocytes (10^12 pcs/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of leukocytes (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of leukocytes (10⁹ pcs/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of hemoglobin (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of hemoglobin (g/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of platelets (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of platelets (10⁹ pcs/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of stab neutrophils (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of stab neutrophils (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of segmented neutrophils (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of segmented neutrophils (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of eosinophils (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of eosinophils (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of basophils (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of basophils (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of monocytes (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of monocytes (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of lymphocytes (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: the content of lymphocytes (in %) is measured. The changes in values between time points are assessed.
Erythrocyte sedimentation rate (ESR) monitoring (as part of a clinical (general) blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a clinical (general) blood test is performed: ESR (in mm/h) is measured. The changes in values between time points are assessed.
Monitoring of the enzyme activity of alanine transaminase (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the enzyme activity of alanine transaminase (in U/l) is measured. The changes in values between time points are assessed.
Monitoring of the enzyme activity of aspartate aminotransferase (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the enzyme activity of aspartate aminotransferase (in U/l) is measured. The changes in values between time points are assessed.
Monitoring of the enzyme activity of lactate dehydrogenase (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the enzyme activity of lactate dehydrogenase (in U/l) is measured. The changes in values between time points are assessed.
Monitoring of the enzyme activity of alkaline phosphatase (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the enzyme activity of alkaline phosphatase (in U/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of B-lipoproteins (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the content of B-lipoproteins (in mmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of cholesterol (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the content of cholesterol (in mmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of total protein (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the content of total protein (in g/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of total bilirubin (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the content of total bilirubin (in µmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of glucose (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the content of glucose (in mmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of creatinine (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the content of creatinine (in µmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of urea (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the content of urea (in mmol/l) is measured. The changes in values between time points are assessed.
Monitoring of thymol test (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the thymol test (in S-H units) is measured. The changes in values between time points are assessed.
Monitoring of the content of C reactive protein (CRP) (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the content of CRP (in mg/ml) is measured. The changes in values between time points are assessed.
Monitoring of the prothrombin index (PTI) (as part of a biochemical blood test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a biochemical blood test is performed: the prothrombin index (in %) is measured. The changes in values between time points are assessed.
Monitoring of urine transparency (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: urine transparency is assessed. The changes in urine transparency between time points are assessed.
Monitoring of the specific gravity of urine (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: the specific gravity of urine is measured. The changes in values between time points are assessed.
Monitoring of the content of protein (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: the content of protein (in g/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of glucose (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: the content of glucose (in mmol / l) is measured. The changes in values between time points are assessed.
Monitoring of the content of leukocytes (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: the content of leukocytes (10⁹/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of erythrocytes (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: the content of erythrocytes (10^12/l) is measured. The changes in values between time points are assessed.
Monitoring of the casts in urine (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: the number of casts in the urine is counted (units in the field of view). The changes in values between time points are assessed.
Monitoring of the salts in urine (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: the number of salt crystals in the urine is counted (crystals per field of view). The changes in values between time points are assessed.
Monitoring of bacteria in urine (as part of a common urine test). | Groups 1, 2, 3: days 0, 5, 14, 21, 30, 60, 90, 180. Group 4: days 0, 5, 12, 21, 28, 37, 67, 97, 187.
  On control days, a common urine test is performed: the number of bacteria in the urine is counted (units in the field of view). The changes in values between time points are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I. Kuzubov, PhD, Principal Investigator — Medical and Sanitary Unit No. 163 (FGBUZ MSCH-163, FMBA Russia)
Locations (1):
- Federal State Budgetary Healthcare Institution - Medical and Sanitary Unit No. 163 of the Federal Medical and Biological Agency (FGBUZ MSCH-163, FMBA Russia), Novosibirsk, Koltsovo, Novosibirsk Region, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yakubitskiy SN, Kolosova IV, Maksyutov RA, Shchelkunov SN. Attenuation of Vaccinia Virus. Acta Naturae. 2015 Oct-Dec;7(4):113-21. PMID 26798498
- [Background] Yakubitskyi SN, Kolosova IV, Maksyutov RA, Shchelkunov SN. Highly immunogenic variant of attenuated vaccinia virus. Dokl Biochem Biophys. 2016;466:35-8. doi: 10.1134/S1607672916010105. Epub 2016 Mar 31. PMID 27025484
- [Background] Maksyutov RA, Yakubitskyi SN, Kolosova IV, Shchelkunov SN. Comparing New-Generation Candidate Vaccines against Human Orthopoxvirus Infections. Acta Naturae. 2017 Apr-Jun;9(2):88-93. PMID 28740731
- [Background] Olson VA, Shchelkunov SN. Are We Prepared in Case of a Possible Smallpox-Like Disease Emergence? Viruses. 2017 Aug 27;9(9):242. doi: 10.3390/v9090242. PMID 32962316
- [Background] Shchelkunova GA, Shchelkunov SN. 40 Years without Smallpox. Acta Naturae. 2017 Oct-Dec;9(4):4-12. PMID 29340212
- [Background] Shchelkunov SN, Shchelkunova GA. [We should be prepared to smallpox re-emergence.]. Vopr Virusol. 2019;64(5):206-214. doi: 10.36233/0507-4088-2019-64-5-206-214. Russian. PMID 32167685
- [Background] Maksyutov RA, Yakubitskiy SN, Kolosova IV, Tregubchak TV, Shvalov AN, Gavrilova EV, Shchelkunov SN. Genome stability of the vaccine strain VACDelta6. Vavilovskii Zhurnal Genet Selektsii. 2022 Jul;26(4):394-401. doi: 10.18699/VJGB-22-48. PMID 35903306
- [Background] Shchelkunov SN, Shchelkunova GA. Genes that Control Vaccinia Virus Immunogenicity. Acta Naturae. 2020 Jan-Mar;12(1):33-41. doi: 10.32607/actanaturae.10935. PMID 32477596
- [Background] Marennikova SS, Shchelkunov SN. Orthopoxviruses pathogenic for humans (monograph). KMK Scientific Press Ltd.1998; 386 p. (in Russian).
- [Background] Kolosova IV, Babkina IN, Yakubitsky SN, Maksyutov RA, Safronov PF, Shchelkunov SN. Recombinant strain L-IVP 1421ABJCN of vaccinia virus with deleted virulence genes A56R, B8R, J2R, C3L, N1L to obtain a live cell-based attenuated vaccine against smallpox and other orthopoxviruses pathogenic to humans. RF Patent No. 2588388, priority 20.04.2015 (in Russian)
- [Background] Yakubitsky SN, Kolosova IV, Maksyutov RA, Shchelkunov SN. Recombinant strain VACΔ6 of vaccinia virus with deleted virulence genes C3L, N1L, J2R, A35R, A56R, B8R for obtaining a live cell-based attenuated vaccine against smallpox and other human orthopoxvirus infections. RF Patent No. 2621868, priority 24.06.2016 (in Russian).